CLINICAL TRIAL: NCT01653444
Title: Multicenter and Dose Escalation Phase 1 Study to Evaluate the Safety and Exploratory Efficacy of GC1119(Recombinant Human α-galactosidase A) for Enzyme Replacement Therapy in Fabry Disease Patients
Brief Title: Evaluate the Safety and Exploratory Efficacy of GC1119
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC1119_P1
Record Dates: First submitted 2012-07-24; First posted 2012-07-31 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GC1119 0.5 mg/kg (Experimental): 0.5 mg/kg biweekly
  Interventions: Drug: GC1119
- GC1119 1.0 mg/kg (Experimental): 1.0 mg/kg biweekly
  Interventions: Drug: GC1119

INTERVENTIONS:
Drug: GC1119 — biweekly, IV infusion

SUMMARY:
The purpose of this study is to evaluate the safety and exploratory efficacy of GC1119 (recombinant human α-galactosidase A) for enzyme replacement therapy in Fabry disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a current diagnosis of Fabry's disease
* Plasma α-gal activity of ≤ 1.5mnol/hr/ml and have a mutation in α-galactosidase A gene
* Males ≥ 16 years old
* Subjects capable of performing this clinical trial in an appropriate manner
* Informed consent form voluntarily signed by the subject(or his legally acceptable representative if the subject is under 20 years old) to participation in the study
* Agreement to contraception during the study period

Exclusion Criteria:

* Serum creatinine > 2.5mg/dl
* Subjects have a plan to kidney transplantation
* Subjects have undergone kidney transplantation
* Subjects are currently on dialysis
* Subjects have a clinically significant organic disease(cardiovascular, hepatic, pulmonary, neurologic, or renal disease)that in the opinion of the investigator would preclude participation in the trial
* Known life-threatening hypersensitivity(anaphylactic reaction) to α-galactosidase
* Treatment with another investigational product within 30days from the administration of study drug dosing or plans to be treated with another investigational product during the study period
* Known hypersensitivity to any of the ingredients of study drug(including excipients)
* Subjects need the medication of prohibited drug
* Alcoholism or drug addiction

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 10weeks

SECONDARY OUTCOMES:
change and %change of Plasma GL-3 concentration | baseline and 10weeks
The ratio of subjects whose plasma GL-3 values are within reference range | 10weeks
change and %change of urine GL-3 concentration | baseline and 10weeks
change and %change of kidney function | baseline and 10weeks
change and %change of kidney size | baseline and 10weeks
change and %change of heart size | baseline and 10weeks
change of results of cornial opacity examination | baseline and 10weeks
change of scores that are measured by pain questionnaire | baseline and 10weeks

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Asan Medical Center, Songpa-gu, Seoul
  - Soon Cung Hyang University Hospital, Yongsan-gu, Seoul
  - Ajou University School of Medicine, Yeongtong-gu, Suwon

IPD SHARING:
Plan to Share IPD: No